CLINICAL TRIAL: NCT00395434
Title: OXC4P1-105: A Phase I Study of the Safety, Tolerability, and Antitumor Activity of Escalating Doses of Combretastatin A4 Phosphate Given in Combination With Bevacizumab to Subjects With Advanced Solid Tumors
Brief Title: Safety Study of Increasing Doses of Combretastatin in Combination With Bevacizumab (Avastin) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mateon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OXC4P1-105
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Last update posted 2011-10-31 (Estimated); Status verified 2011-10

CONDITIONS: Tumors
Keywords: Advanced Solid Tumors; Advanced Solid Tumours; Advanced Solid Tumor; Advanced Solid Tumour; Advanced; Malignant; Solid; Tumors; Tumours; Tumor; Tumour; Cancer; Malignant Solid Tumors; Malignant Solid Tumours; Malignant Solid Tumor; Malignant Solid Tumour; Metastatic Cancer; Metastatic Disease; Advanced Cancer; Vascular Disrupting Agent; Anti-angiogenesis agent; Phase 1
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — fosbretabulin; Bevacizumab

INTERVENTIONS:
Drug: Combretastatin A4 Phosphate (CA4P)
Drug: Bevacizumab (Avastin)

SUMMARY:
The purpose of this study is to determine the safety and tolerability of three dose levels of combretastatin A4 phosphate (CA4P) given intravenously (IV) in combination with bevacizumab every 14 days in patients with advanced solid tumors. The maximum tolerated dose will be defined if it is at one of the three dose levels under study.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically or cytologically confirmed malignant solid tumors that have failed standard therapy or for which no life prolonging treatment exists
2. Measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria
3. At least 4 weeks since any prior immunotherapy, chemotherapy or radiation therapy prior to first dose of study drug (six weeks for therapy known to be associated with delayed toxicity such as nitrosoureas or mitomycin-C)
4. Age > or = to 18 years old
5. Adequate bone marrow function:

   1. absolute granulocyte count (neutrophils and bands) > or = to 1500 cells/mm3;
   2. platelet count > or = to 100,000 cells/mm3;
   3. hemoglobin > or = to 9 g/dL.
6. Adequate renal function (glomerular filtration calculated by Cockcroft/Gault formula or measure urine creatinine clearance > or = to 50 mL/minute)
7. Adequate hepatic function:

   1. bilirubin less than or = to 1.5 mg/dL;
   2. aspartate transaminase (AST) and alanine transaminase (ALT) less than or = to 2.5 times the institutional upper limit of normal (ULN) (or less than or = to 5 times ULN if liver metastases are present).
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
9. Life expectancy of > or = to 12 weeks
10. Written, signed, dated, and witnessed (if applicable as per International Conference on Harmonization [ICH] guidelines) Independent Ethics Committee (IEC) approved informed consent form before any study specific screening procedures are performed
11. Fertile subjects must abstain from sexual intercourse or use effective birth control.
12. All women of child bearing potential (WOCBP) must have a negative serum pregnancy test within 72 hours of first dose.

Exclusion Criteria:

1. Contraindications, allergies or sensitivity to the use of the study medications or any other products required for participation in this study (i.e. contrast agents)
2. Presence of central nervous system (CNS) metastases
3. Diagnosed squamous non-small cell lung cancer (NSCLC)
4. History of gastrointestinal perforations
5. Surgery within 28 days of screening visit or a surgical incision that is not fully healed. Any surgery planned during the study period.
6. Proteinuria >1 g/24 hours by 24 hour urine collection (perform 24 hour urine collection if > 1+ on dipstick)
7. Recent hemoptysis (occurrence within the past 3 months)
8. Prior therapy with CA4P or bevacizumab, or other agents which target vascular endothelial growth factor (VEGF) or VEGFR signaling such as Sorafenib and Sutent
9. Prior radiation involving > 30% of the bone marrow
10. Radical radiotherapy to the thorax or abdomen at any time or post-operative radical radiotherapy to the pelvis. Palliative radiotherapy treatments are acceptable. Subjects with rectal primaries who have received pre-operative pelvic radiotherapy or chemoradiation are eligible if the small bowel was mobile and not stuck to the tumor.
11. Active autoimmune disorder(s)
12. Immunocompromised, including subjects known to be human immunodeficiency virus (HIV) positive
13. Active infection requiring antibiotic therapy or any other serious intercurrent illness
14. History of angina (stable or severe, even if controlled with medications), myocardial infarction, congestive heart failure (CHF), non-controlled atrial arrhythmias or clinically significant arrhythmias including conduction abnormality, nodal junctional arrhythmias and dysrhythmias, sinus bradycardia or tachycardia, supraventricular arrhythmias, atrial fibrillation or flutter, syncope or vasovagal episodes
15. Electrocardiogram (ECG) with evidence of prior myocardial infarction (e.g., significant Q waves), QTc > 450 msec or other clinically significant abnormalities
16. Taking any drug(s) known to prolong the QTc interval, which cannot be interrupted for at least four days during each treatment cycle.
17. Known significant heart wall abnormality or heart muscle damage as evidenced on multiple-gated acquisition (MUGA) scan or echocardiogram (this is not a required screening investigation)
18. Uncontrolled hypertension (defined as blood pressure consistently greater than 150/100 irrespective of medication). Or controlled hypertension requiring use of > 2 classes of anti-hypertensives.
19. Uncontrolled hypokalemia and/or hypomagnesemia
20. Symptomatic peripheral vascular disease or cerebrovascular disease
21. Psychiatric disorders or other conditions rendering subjects incapable of complying with the requirements of the protocol
22. Receiving concurrent hormonal therapy with the exception of gonadotropin-releasing hormone (GnRH) agonists in subjects with hormone refractory prostate cancer, hormone replacement therapy (HRT), oral contraceptives, and megestrol acetate used for anorexia/cachexia
23. Receiving anticoagulation with warfarin, heparin or low molecular weight heparin other than low dose (1 mg) warfarin for maintenance of central line patency
24. Women who are currently pregnant, nursing, or planning a pregnancy; or women who have a positive pregnancy test.
25. Receiving concurrent antineoplastic therapy (radiation therapy, cytotoxic or biologic therapy)
26. Participation in an investigational drug or device trial within 30 days of entering the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-09; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of the combination therapy assessed by analysis of adverse events
safety and tolerability of the combination therapy assessed by analysis of laboratory tests
safety and tolerability of the combination therapy assessed by analysis of other assessments within the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Paul Nathan, MD, Principal Investigator — Mount Vernon Hospital; Hillori Connors, MS, Study Director — Mateon Therapeutics; Peter Harris, MD, Study Director — Mateon Therapeutics
Locations (2):
- United Kingdom (2):
  - Mount Vernon Hospital, Northwood, Middlesex
  - Royal Marsden Hospital, Sutton, Surrey